CLINICAL TRIAL: NCT02289092
Title: Testing the Efficacy of an Ecological Approach to Family Intervention and Treatment During Early Elementary School to Prevent Problem Behavior and Improve Academic Outcomes
Brief Title: The Positive Family Support Project - Partnering With Families for a Successful Transition to School
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of Oregon (Other)
Responsible Party: Principal Investigator, Beth Stormshak, Principal Investigator, University of Oregon
Allocation: Randomized | Model: Single Group | Masking: None | Purpose: Prevention
Other Study IDs: 05142014.022
Record Dates: First submitted 2014-10-14; First posted 2014-11-13 (Estimated); Last update posted 2022-06-21 (Actual); Status verified 2022-06

CONDITIONS: Achievement

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- Family Check-Up Intervention (Experimental): Prior to the feedback session, trained clinicians will observe family interactions by reviewing the video-taped observations and questionnaires filled out by parents. Therapists then use this data to inform the intervention process and provide feedback to parents based on norms for this age period. Feedback sessions will include a discussion of goal attainment and plans to achieve goals, with specific attention to the parent's role in supporting positive behavior. Options for obtaining goals are based on the literature about empirically supported interventions for this age group and include (a) periodic follow-up and support, (b) brief support for change on a specific topic, and (c) community referral (e.g., substance abuse referral; domestic violence referral; referral for individual therapy for depression; referral for family therapy and support for families in conflict).
  Interventions: Behavioral: Family Check-Up
- Control (No Intervention): Control families will receive services as usual that are being provided to the families within their school

INTERVENTIONS:
Behavioral: Family Check-Up — Parents fill out questionnaires about their child and families and then participate in a videotaped interaction with their child. Clinicians then observe the video and analyze the questionnaires to establish family needs based on supports, stress, parenting, values, and strengths. Therapists then use this information to inform the intervention process and provide feedback to families with the use of motivational interviewing. parents identify goals for parenting and/or child behavior and to connect them with resources when needed. Feedback includes a discussion of goal attainment and plans to achieve goals. Goal achievement includes options such as (a) periodic follow-up and support, (b) brief support for change on a specific topic, and (c) community referral (e.g., substance abuse referral; domestic violence referral; referral for individual therapy for depression; referral for family therapy and support for families in conflict).
  Other Names: Positive Family Support
  Arms: Family Check-Up Intervention

SUMMARY:
The Positive Family Support Project seeks to understand some of the factors that increase success for children in early elementary school, such as positive family support at home. This study will inform us on ways to help children learn and succeed in school.

DETAILED DESCRIPTION:
The transition to elementary school is a critical time for the development of key skills that are necessary for school success, including sustained attention, self-regulation, initiating and sustaining successful peer relationships, and academic competence. Parent support at home, such as positive parenting and support for learning, is associated with school readiness indicators that predict successful adaptation to the school context. For many children at risk for poor developmental outcomes this transition can be difficult and may lead to early academic problems, which in turn may define a trajectory that culminates in more severe forms of problem behavior and learning difficulties. The purpose of this study is to evaluate the efficacy of implementing the Family Check-Up (FCU), a school-based, ecological approach to family intervention, during the transition into elementary school.

ELIGIBILITY:
Inclusion Criteria: 700 Kindergarten children and their families entering Kindergarten in the Clackamas School District in 2014 and 2015 -

Exclusion Criteria:

-

Sex: All | Healthy Volunteers: Yes
Age Groups: Child, Adult, Older Adult
Enrollment: 848 (Actual)
Dates: Start 2014-09 (Actual); Primary Completion 2019-06-30 (Actual); Study Completion 2019-06-30 (Actual)

PRIMARY OUTCOMES:
Change in parenting skills measured by standardized questionnaires | Up to 3 years
  Change in parenting skills for parents participating in the intervention arm measured by standardized questionnaires
Change in child self-regulation and behavioral control measured by standardized questionnaires | Up to 3 years
  Change in child self-regulation in the classroom for children participating in the intervention arm in comparison to children participating in the control arm measured by standardized questionnaires
Increase chances for child school success as measured by early literacy standardized testing scores | Up to 3 years
  Increase chances for success in school for children participating in the intervention arm in comparison to children participating in the control arm as measured by early literacy standardized testing scores
Increase positive child social relationships as measured by standardized questionnaires | Up to 3 years
  Increase positive social relationships in child participating in the intervention arm in comparison with children in the control arm as measured by standardized questionnaires

SECONDARY OUTCOMES:
Decrease in family stress/hardship as measured by standardized questionnaires | Up to 3 years
  Decrease in family stress and or hardship for families participating in the intervention arm as measured by standardized questionnaires

CONTACTS AND LOCATIONS:
Locations (1):
- University of Oregon Child and Family Center, Eugene, Oregon, United States

REFERENCES:
- [Derived] Hails KA, McWhirter AC, Garbacz SA, DeGarmo D, Caruthers AS, Stormshak EA, McIntyre LL. Parenting self-efficacy in relation to the family check-up's effect on elementary school children's behavior. J Fam Psychol. 2024 Sep;38(6):858-868. doi: 10.1037/fam0001237. Epub 2024 May 23. PMID 38780604
- [Derived] Flack CE, Garbacz SA, Stormshak EA, McIntyre LL. A longitudinal study of home-based involvement and dyadic adjustment during the transition to early elementary school. Sch Psychol. 2023 Sep;38(5):287-293. doi: 10.1037/spq0000543. Epub 2023 Mar 30. PMID 36996236
- [Derived] Resnik F, Garbacz SA, Stormshak EA, McIntyre LL. Family-centered prevention to enhance proactive parenting and parental self-efficacy during early elementary school. J Fam Psychol. 2023 Apr;37(3):380-387. doi: 10.1037/fam0001050. Epub 2023 Jan 9. PMID 36622726
- [Derived] Stormshak EA, DeGarmo D, Garbacz SA, McIntyre LL, Caruthers A. Using Motivational Interviewing to Improve Parenting Skills and Prevent Problem Behavior During the Transition to Kindergarten. Prev Sci. 2021 Aug;22(6):747-757. doi: 10.1007/s11121-020-01102-w. PMID 32036553
- [Derived] Stormshak EA, McIntyre LL, Garbacz SA, Kosty DB. Family-centered prevention to enhance parenting skills during the transition to elementary school: A randomized trial. J Fam Psychol. 2020 Feb;34(1):122-127. doi: 10.1037/fam0000570. Epub 2019 Jul 18. PMID 31318264